CLINICAL TRIAL: NCT06402292
Title: Outcomes of Surgical Treatment of Osteoarticular Infections Using Bioactive Bone Substitute Impregnated With Antibiotics: Prospective Study
Brief Title: Surgical Treatment of Osteoarticular Infections Using Bioactive Bone Substitute
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, GUILHERME GUADAGNINI FALOTICO, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FALOTICO
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Osteomyelitis; Infections; Fracture; Antibiotics
Keywords: infection; osteomyelitis; fracture; local antibiotics
MeSH Terms: conditions — Osteomyelitis; Infections; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATIENTS WITH FRACTURE-RELATED INFECTION (FRI GROUP) (Experimental): USE OF LOCAL ANTIBIOTICS WITH PEROSSAL
  Interventions: Procedure: OSTEOMYELITIS SURGICAL TREATMENT WITH LOCAL ANTIBIOTICS AND PEROSSAL

INTERVENTIONS:
Procedure: OSTEOMYELITIS SURGICAL TREATMENT WITH LOCAL ANTIBIOTICS AND PEROSSAL — 25 PATIENTS WITH FRI WILL BE SURGICALLY TREAT WITH DESBRIDMENT AND PEROSSAL WITH ANTIBIOTCS

SUMMARY:
This prospective research project aims to evaluate the effectiveness and clinical outcomes of utilizing antibiotic-impregnated bioactive bone substitute (PerOssal®) in the surgical management of osteoarticular infections. Osteoarticular infections pose significant challenges in orthopaedic surgery due to the risk of persistent infection, bone loss, and functional impairment. Traditional treatment approaches involve extensive debridement followed by systemic antibiotic therapy and bone grafting. However, antibiotic-impregnated bioactive bone substitutes offer a promising alternative by providing local antibiotic delivery and promoting bone regeneration simultaneously. This study will prospectively enrol patients undergoing surgical intervention for osteoarticular infections and assess their clinical outcomes, including infection resolution, bone healing, functional recovery, and complication rates. Comprehensive data collection will include preoperative patient characteristics, intraoperative details, postoperative outcomes, and long-term follow-up assessments. Statistical analyses will be performed to compare outcomes between patients treated with antibiotic-impregnated bioactive bone substitute and those past managed with traditional methods. The findings of this study are expected to contribute valuable insights into the effectivennes and safety of this novel approach, potentially informing future clinical practices and optimizing patient care in the management of osteoarticular infections.

DETAILED DESCRIPTION:
Background:

Osteoarticular infections represent a significant challenge in orthopedic surgery, posing substantial morbidity and potential mortality if not adequately managed. These infections can arise from various sources, including hematogenous spread, contiguous spread from adjacent soft tissue or bone, or direct inoculation during trauma or surgery. Common pathogens associated with osteoarticular infections include Staphylococcus aureus, coagulase-negative staphylococci, Streptococcus species, and gram-negative bacilli, among others.

The management of osteoarticular infections typically involves a combination of surgical intervention and antimicrobial therapy. Surgical treatment aims to achieve complete debridement of infected tissue, removal of necrotic bone, and restoration of skeletal integrity. However, achieving adequate debridement and local antibiotic delivery while preserving bone stock remains a challenge.

Traditional approaches to bone defect management often rely on autografts, allografts, or synthetic bone substitutes. While these methods have demonstrated efficacy in promoting bone healing, they may not address the specific challenges posed by osteoarticular infections, particularly in terms of infection eradication and local antibiotic delivery.

In recent years, there has been growing interest in the use of antibiotic-impregnated bioactive bone substitutes for the management of osteoarticular infections. These materials offer several potential advantages over traditional approaches. Firstly, they provide a scaffold for bone regeneration, promoting osteogenesis and osteoconduction. Secondly, they have the capacity to release antibiotics locally, achieving high concentrations at the site of infection while minimizing systemic exposure and potential adverse effects. Thirdly, they can fill osseous defects and provide structural support, facilitating functional recovery.

The efficacy of antibiotic-impregnated bioactive bone substitutes in the treatment of osteoarticular infections has been investigated in several preclinical and clinical studies. Preclinical studies have demonstrated the ability of these materials to effectively deliver antibiotics, inhibit bacterial growth, and promote bone healing in animal models of osteomyelitis and septic arthritis. Clinical studies have reported promising results, including high rates of infection resolution, bone healing, and functional recovery, with low rates of recurrence and complications.

However, despite these promising findings, there remains a need for further research to evaluate the long-term outcomes and comparative effectiveness of antibiotic-impregnated bioactive bone substitutes in the surgical management of osteoarticular infections. Additionally, questions regarding the optimal selection of antibiotics, the timing and duration of local antibiotic delivery, and the potential for antibiotic resistance warrant investigation.

Therefore, this prospective research project aims to address these gaps in knowledge by evaluating the outcomes of surgical treatment of osteoarticular infections using antibiotic-impregnated bioactive bone substitutes in a well-defined patient population. By systematically assessing clinical outcomes, including infection resolution, bone healing, functional recovery, and complication rates, this study seeks to provide evidence-based insights into the efficacy and safety of this novel approach. Ultimately, the findings of this study may have implications for clinical practice, guiding the optimization of surgical management strategies for osteoarticular infections and improving patient outcomes.

Hypothesis The utilization of antibiotic-impregnated bioactive bone substitute reduces recurrence in patients with osteoarticular infections compared to untreated patients. It presents clinical non-inferiority and decreases hospitalization time in relation to the use of PMMA, as it does not require another surgical procedure for material removal.

Clinical Question:

PICOS Strategy P (Patients): Patients above 12 years old with fracture-related infection (FRI) and indication for surgical treatment.

I (Intervention): Orthopedic surgical treatment with standard local debridement, supplemented with implantation of antibiotic-impregnated bioactive bone substitute (PerOssal®).

C (Control): Retrospective cohort of previously operated patients without the use of local treatment or with the use of antibiotic-loaded PMMA.

O (Outcomes):

Primary: Comparative rate of infection recurrence within 1-year follow-up. Secondary: Pain score, quality of life, overall complications, microbiological profile of infections, duration of systemic antibiotic usage, length of hospital stay.

S (Study): Prospective cohort.

Methods:

This is an observational, prospective, single-center study. The methodology will be guided by the STROBE checklist and the study submitted to the Plataforma Brasil and Ethics Committee. Data will be collected using RedCap® Protocol.

Sample size calculation: For comparison of relative risk between groups, expecting a mean difference of 20% in infection recurrence rate between patients without local antibiotic treatment and patients with local treatment, the expected necessary number of patients is 20. Accounting for a 20% loss to follow-up, the required number of patients in the study will be 25.

Statistical Analysis:

Quantitative Variables:

* T-test and ANOVA for parametric data.
* Mann-Whitney or Kruskal-Wallis tests for non-parametric data.

Qualitative Variables:

- Fischer's exact test.

Relative Risk:

- Cox regression.

Descriptive Values:

- Mean and standard deviation; 95% confidence interval.

Statistical Significance:

- p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

All fracture-related infections (clinical and laboratory/microbiological diagnosis).

Patients > 12 years old.

Surgical treatment with indication for local antibiotic use.

Exclusion Criteria:

Other modalities of musculoskeletal infection (arthroplasties, hematogenous osteomyelitis, septic arthritis, infections related to bone tumors).

Unconfirmed diagnosis of infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Comparative rate of infection recurrence | 1 YEAR

SECONDARY OUTCOMES:
Pain score using numeric pain scale (0 - no pain; 10 - worst pain) | 6,12, 24, 48 WEEKS
QUALITY OF LIFE USING EuroQol-5D (EQ-5D) | 6,12, 24, 48 WEEKS
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
General complications (other than infection recurrence) | 6,12, 24, 48 WEEKS
  clinical issues (thrombosis, pneumonia, urinary infection, cardic descompensation); shock; hemorrhage; blood transfusion; neurovascular injury.
Microbiological profile of infections | up to 1 week
  Detailed description of microorganisms found in tissue cultures and sonication results (agent group, antimicrobial resistance profile, antibiogram)
Duration of systemic antibiotic usage | up to 12 weeks
Length of hospital stay | through study completion, an average of 1 year
  The length of hospitalization for each patient will be defined at the end of the study (it will include the time of all hospitalizations in patients with eventual recurrence and the need for new surgical approaches)

CONTACTS AND LOCATIONS:
Overall Officials: GUILHERME FALOTICO, PhD, Principal Investigator — PROFESSOR

IPD SHARING:
Plan to Share IPD: No